CLINICAL TRIAL: NCT03087864
Title: PDL-1 Targeting in Resectable Oesophageal Cancer: a Phase II Feasibility Study of Atezolizumab and Chemoradiation.
Brief Title: PDL-1 Targeting in Resectable Oesophageal Cancer
Acronym: PERFECT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: UMC Utrecht (Other)
Responsible Party: Principal Investigator, H.W.M. van Laarhoven, Prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016_325
Record Dates: First submitted 2017-03-14; First posted 2017-03-23 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Esophageal Cancer, Stage II; Esophageal Cancer Stage III
Keywords: esophageal cancer; PD-L1 inhibition; chemoradiation
MeSH Terms: conditions — Esophageal Neoplasms | interventions — atezolizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atezolizumab and Chemoradiation (Experimental): Atezolizumab 1200 mg i.v. day 1-22-43-64-85 Carboplatin AUC = 2 i.v day 1-8-15-22-29 Paclitaxel 50 mg/m2 i.v day 1-8-15-22-29 Radiotherapy 23 x 1.8 Gy
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiotherapy 23 x 1.8 Gy

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1200 mg i.v. day 1-22-43-64-85
Drug: Carboplatin — Chemotherapy
Drug: Paclitaxel — Chemotherapy
Radiation: Radiotherapy 23 x 1.8 Gy — Radiotherapy

SUMMARY:
Objectives The primary objective of this study is to assess the feasibility of preoperative treatment with atezolizumab combined with preoperative chemoradiation (carboplatin, paclitaxel and radiation) in terms of completion of treatment with atezolizumab.

DETAILED DESCRIPTION:
Objectives The primary objective of the study of this study is to assess the feasibility of preoperative treatment with atezolizumab combined with preoperative chemoradiation (carboplatin, paclitaxel and radiation) in terms of completion of treatment with atezolizumab.

Secondary objectives are:

* To assess toxicities of atezolizumab alone and in combination with chemoradiation.
* To assess completion of chemotherapy and radiation treatment
* To assess withdrawal rate from surgery
* To assess post-operative complications.
* To assess pathological response.
* To assess R0 resection rate.
* To assess the relation between gut microbiota composition and response.
* To assess the relation between gut microbiota composition and toxicity.

Explorative objectives are:

To perform exploratory biomarker analyses from tumor tissue and blood-derived samples and correlate with safety and clinical outcome. Biomarker analyses include (but are not limited to):

* Expression of PD-1, PD-L1 and FOXP3, presence of tumor infiltrating CD8+/CD4+ cytotoxic/helper T lymphocytes, IFNγ expression, presence of tumor macrophages, STAT3 and STAT6 expression, MHC classI, MHC class II, EBV and MSI status on tumor tissue.
* RNA sequencing and whole exome sequencing to develop a predictive profile for response to treatment.
* Analysis of ctDNA extracted from plasma of patients at four time points (baseline, directly after chemoradiation, at surgery and 3 months after surgery) and analyzed using Ion Torrent Next Generation sequence technology as a non-invasive marker for response to treatment.
* Analysis of peripheral blood mononuclear cells (PBMCs) extracted from whole blood of patients at three time points ((baseline, directly after chemoradiation, at surgery) )
* Duodenal biopsy and morning faeces sample analysis as predictor of response will be done by HIT Chip flora mapping, an established sensitive RT-qPCR method which is developed for exact and sensitive enumeration of bacterial population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the esophagus or gastro esophageal junction.
* Surgical resectable (<T4b, N0 or N+, M0), as determined by Endoscopic Ultra Sound (EUS) and CT scan of neck, thorax and abdomen. Tumors that cannot be passed with an endoscope for endoscopic ultrasound are eligible if all other criteria are fulfilled.
* T1N+ tumors are eligible.
* Tumor length longitudinal ≤ 10 cm; if larger than 10 cm, inclusion should be discussed with the principal investigator.
* If the tumor extends below the gastroesophageal (GE) junction into the proximal stomach, the bulk of the tumor must involve the esophagus or GE junction.
* Age ≥ 18.
* ECOG performance status 0 or 1 (cf. Appendix A).
* Adequate hematological, renal and hepatic functions defined as:

  * neutrophiles ≥ 1.5 x 109/L
  * platelets ≥ 100 x 109/L
  * hemoglobin ≥ 5.6 mmol
  * total bilirubin ≤ 1.5 x upper normal limit
  * creatinine clearance (Cockroft) > 60 ml/min
* Written, voluntary informed consent
* Patients must be accessible to follow up and management in the treatment center

Exclusion Criteria:

* Past or current history of malignancy other than entry diagnosis interfering with prognosis of esophageal cancer.
* Invasion of the tracheobronchial tree or presence of tracheoesophageal fistula.
* T1N0 tumors or in situ carcinoma.
* Pregnancy (positive serum pregnancy test), planning to become pregnant, and lactation.
* Patient (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment.
* Previous chemotherapy, radiotherapy, and/or treatment with checkpoint inhibitors.
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) precluding major surgery.
* Pulmonary fibrosis and/or severely impaired lung function precluding major surgery.
* Pre-existing motor or sensory neurotoxicity greater than WHO grade 1.
* Serious underlying medical condition which would impair the ability of the patient to receive the planned treatment, including prior allergic reactions to drugs containing Cremophor, such as teniposide or cyclosporine.
* Dementia or altered mental status that would prohibit the understanding and giving of informed consent
* Inadequate caloric- and/or fluid intake despite consultation of a dietician and/or tube feeding.
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine for patients with a history of autoimmune-related hypothyroidism, insulin for patients with type 1 diabetes mellitus, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Patients with vitiligo with dermatological manifestations only are eligible to enter the study.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (>10 mg/day prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy which has not resolved 3 days (simple infection such as cystitis) to 7 days (severe infection such as pyelonephritis) prior to the first dose of trial treatment.
* Patients with prior allogeneic stem cell or solid organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
feasibility defined as percentage completion of treatment with atezolizumab. | up to 3 months
  The primary endpoint is feasibility defined as percentage completion of treatment with atezolizumab

SECONDARY OUTCOMES:
Incidence and severity of toxicity | up to 3 months
  Incidence and severity of toxicity defined to CTCAE v4.03 and Radiation Oncology Group (RTOG) criteria.
Percentage completion of chemotherapy and radiation treatment | up to 3 months
  Percentage completion of chemotherapy and radiation treatment
Percentage withdrawal rate from surgery due to atezolizumab related complications | up to 3 months
  Percentage withdrawal rate from surgery due to atezolizumab related complications
Percentage delay of surgery due to atezolizumab related complications | up to 3 months
  Percentage delay of surgery due to atezolizumab related complications
Incidence and severity of post-operative complications to the Dindo classification | up to 3 months
  Incidence and severity of post-operative complications to the Dindo classification
Pathological response according to the Mandard criteria | up to 3 months
  Pathological response according to the Mandard criteria
R0 resection rate. | up to 3 months
  R0 resection rate.
Progression free survival | up to 3 months
  Progression free survival
Overall survival | up to 3 months
  Overall survival

OTHER OUTCOMES:
Potential biomarker development based on assessment of tumour biopsies, blood- and faecal samples and the proposed mechanism of action of study drugs. | up to 3 months
  Potential biomarker development based on assessment of tumour biopsies, blood- and faecal samples and the proposed mechanism of action of study drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke WM van Laarhoven, Prof. dr., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Medical Oncology, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van den Ende T, Ezdoglian A, Baas LM, Bakker J, Lougheed SM, Harrasser M, Waasdorp C, van Berge Henegouwen MI, Hulshof MCCM, Haj Mohammad N, van Hillegersberg R, Mook S, van der Laken CJ, van Grieken NCT, Derks S, Bijlsma MF, van Laarhoven HWM, de Gruijl TD. Longitudinal immune monitoring of patients with resectable esophageal adenocarcinoma treated with Neoadjuvant PD-L1 checkpoint inhibition. Oncoimmunology. 2023 Jul 17;12(1):2233403. doi: 10.1080/2162402X.2023.2233403. eCollection 2023. PMID 37470057
- [Derived] van den Ende T, Menting SP, Ambarus CA, van Oijen MGH, van Laarhoven HWM. Cutaneous Toxicity After Chemoradiotherapy and PD-L1 Inhibition in Two Patients with Esophageal Adenocarcinoma: More than Meets the Eye. Oncologist. 2019 Apr;24(4):e149-e153. doi: 10.1634/theoncologist.2018-0674. Epub 2019 Mar 22. PMID 30902915